CLINICAL TRIAL: NCT07064629
Title: DigiWell - Relaxation Breathing in Virtual Reality Using Biofeedback
Brief Title: Training of Relaxation Breathing in Virtual Reality Using Biofeedback: Comparison Study
Acronym: VRrelaxBF
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health, Czech Republic (Other)
Responsible Party: Principal Investigator, Iveta Fajnerová, Supervisor, National Institute of Mental Health, Czech Republic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: DigiWell_Relax_01; CZ.02.01.01/00/22_008/0004583 (Other Grant/Funding Number: MEYS, Programme Johannes Amos Comenius co-financed by the European Union)
Record Dates: First submitted 2025-06-13; First posted 2025-07-15 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Relaxation; Anxiety Disorders; Biofeedback Training
Keywords: Virtual reality; relaxation; breathing techniques; anxiety disorders; biofeedback
MeSH Terms: conditions — Anxiety Disorders | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality relaxation breathing with/without biofeedback (Experimental): Intervention group 1: use of VR application for relaxation breathing in the first two sessions with biofeedback, followed by two sessions without biofeedback.
  Interventions: Behavioral: Relaxation in virtual reality with biofeedback.; Behavioral: Relaxation in virtual reality without biofeedback
- Virtual reality relaxation breathing without/with biofeedback (Active Comparator): Intervention group 2: use of VR application for relaxation breathing in the first two sessions without biofeedback, followed by two sessions with biofeedback.
  Interventions: Behavioral: Relaxation in virtual reality with biofeedback.; Behavioral: Relaxation in virtual reality without biofeedback

INTERVENTIONS:
Behavioral: Relaxation in virtual reality with biofeedback. — In this intervention, biofeedback is provided based on the respiratory rate measured by a Vernier Go respiration belt. This belt sends signals (respiratory effort) to the application that calculates the level of synchronisation and gives the visual biofeedback in two forms: 1) a deer simultanously breathing with the participant (realtime biofeedback, present in the initial phase only), 2) a growing tree - if breathing is regulated following a given rhytm, a growing tree is giving the targeted biofeedback.
  Other Names: withBF
Behavioral: Relaxation in virtual reality without biofeedback — In this control intervention, participants' respiratory rate is still being measured by the respiratory belt VernierGo; however, they are not receiving any visual biofeedback inside the virtual relaxation application (no deer is present, the tree is constantly growing regardless of the breathing pattern of the participant).
  Other Names: withoutBF

SUMMARY:
This study aims to evaluate the effectiveness of a VR-based relaxation breathing training with biofeedback compared to a non-biofeedback version in patients with anxiety disorders. The randomized controlled trial will include at least 30 participants (15 per group) diagnosed with an anxiety disorder (DSM-5 or ICD-10 criteria). The intervention will use BreezeTerraVR, a custom-built virtual reality (VR) application developed by VR research center team members at NIMH. This app provides training in deep relaxation breathing technique with or without biofeedback (BF - visual elements reflecting real-time breathing patterns measured via breathing belt) in a virtual nature environment. This study compares two subgroups of anxiety patients, both completing four 20-minute intervention sessions, two sessions with BF and two without BF (in randomized order).

This study will assess the feasibility of the VR intervention, estimate effect sizes, and provide preliminary insights into its impact on relaxation training in individuals with anxiety disorders.

This study is funded by the European Union's co-financed project "Research of Excellence on Digital Technologies and Wellbeing CZ.02.01.01/00/22_008/0004583."

DETAILED DESCRIPTION:
This study evaluates the efficacy of a virtual reality (VR)-based relaxation intervention incorporating real-time respiratory biofeedback, delivered via a standalone Meta Quest 2 headset. This study uses a randomized crossover design in which all participants undergo two sessions of virtual reality (VR) relaxation with biofeedback, followed by two sessions without biofeedback, or vice versa. The order of conditions is randomized to control for order effects. The randomization is done via an online randomization tool.

The intervention utilizes a custom-developed application-BreezeTerraVR-designed by the research team at the Center for Virtual Reality Research in Mental Health and Neuroscience, part of the National Institute of Mental Health (NIMH), Czech Republic. BreezeTerraVR is a structured and modifiable VR application specifically built to facilitate training in slow-paced, rhythmic breathing, allowing flexible adjustments to the inhalation, exhalation, and breath-hold phases according to research needs or participant abilities.

The virtual environment represents a calming natural meadow, surrounded by trees. Participants are immersed in this nature scene and guided to practice square (box) breathing, consisting of 4 seconds inhale, 4 seconds hold, 4 seconds exhale, and 4 seconds hold. The target breathing rhythm is visualized through a colored mist moving between two concentric mushroom-shaped circles in the visual field.

Two distinct biofeedback modalities are integrated into the VR experience for the intervention condition with BF:

1. Real-time biofeedback is represented by an animated deer walking in front of the user. The deer's exhalation is visualized with visible steam from its nostrils, mirroring the participant's actual breathing rhythm as measured by a Go Direct® Respiration Belt (Vernier).
2. Targeted biofeedback is represented by a tree located at the center of the mushroom circle. This tree dynamically grows or shrinks depending on how closely the participant's breathing matches the set rhythm. The feedback difficulty can be adjusted to four levels (0-3), the study protocol applied Level 2 (moderate): Accurate rhythm required for growth; the tree can shrink if the breathing is out of a given rhythm.

In the control condition (Intervention 2), participants engage with the same VR environment and breathing pattern but without biofeedback elements: the deer and the tree are not present. Visual and auditory guidance is still provided via the mist and voice instructions, but there is no adaptive feedback.

All recruited participants sign an Informed consent to participate in the study.

The study duration is three weeks with 4 relaxation sessions in total. The participants complete two VR relaxations per week (e.g.Tuesdays and Thursdays). After the first week of interventions, a one-week break is implemented. The third week the same protocol with two additional sessions is completed. This means the participants complete one of the interventions (conditions) in the first week and the other intervention in the third week.

Each study session takes no longer than 25 minutes per participant. Each of the 4 sessions includes a pre-intervention baseline assessment, a standardized VR breathing session (5 minutes duration) with 3 additional minutes before and 3 minutes after the relaxation spent in the VR environment to measure the pre/post respiratory rate, and a post-intervention assessment. The participants complete the given questionnaires on tablets or computers.

The primary outcomes measured before and after each session include:

* Subjective change in anxiety
* Self-reported relaxation state
* Objective physiological change in respiratory rate (measured for 3 minutes before and after the relaxation).

Secondary outcomes completed only once, immediately after the final Session 4, include the sense of presence and cybersickness measures.

Data will be analyzed using appropriate statistical methods based on sample size and distribution characteristics. Parametric or non-parametric tests (e.g., t-tests, ANOVA, LLM, Mann-Whitney U, or Wilcoxon signed-rank tests) will be used to evaluate within- and between-group differences in anxiety reduction, relaxation level, and physiological measures. Additional analyses may explore interactions between biofeedback accuracy, presence, and outcome effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* patients with Anxiety disorders

Exclusion Criteria:

* severe neurological disease (e.g. epilepsia)
* psychiatric disorders other then Anxiety disorder
* serious somatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | - baseline/pre-intervention (for 3 minutes) - during the intervention (for 5 minutes) - immediately after the intervention (for 3 minutes)
  Data from the breathing pattern (respiration effort and respiration rate) measured at the baseline before the beginning of the relaxation, during the relaxation, and a period after the relaxation. The measure is repeated in each session 1-4.
Acute symptoms of anxiety | - baseline/pre-intervention (before each session) - and immediately after the intervention (after each session)
  Using the short version of the State-Trait Anxiety Inventory (STAI-6) questionnaire, measures of acute anxiety symptoms before and after each relaxation session (sessions 1-4). Higher scores indicate higher anxiety. The lowest possible score is 6 (minimum anxiety), and the highest is 24 (maximum anxiety).
State of relaxation | - Baseline/pre-intervention (each session) - and immediately after the intervention (each session).
  With the Relaxation State Questionnaire (RSQ), measured before and after each relaxation session (sessions 1-4). Higher scores imply higher subjective perception of being relaxed. The lowest possible score is 10 (the least relaxed), and the highest is 50 (maximum relaxation).

SECONDARY OUTCOMES:
Simulator sickness | Immediately after finishing the final intervention session (Session 4).
  With the Simulation Sickness Questionnaire (SSQ), the potential cybersickness symptoms are measured. Higher scores indicate higher cybersickness. The total score is the sum of subscores from all 16 items and can range from 0 (no symptoms) to 48 (highest symptom intensity).
Sense of presence | Immediately after finishing the final intervention session (Session 4).
  With the iGroup Presence Questionnaire (IPQ), we measure the perceived ability to be immersed in the virtual environment. The total IPQ score is calculated by averaging the responses to all 14 items on the questionnaire. The lowest possible mean score is -3, while the highest mean score is 3. Higher scores indicate a higher sense of presence.

CONTACTS AND LOCATIONS:
Overall Officials: Iveta Fajnerova, PhD., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institute of Mental Health, Klecany, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: Yes
IPD (primary outcome measures) that underlie results in a publication.
Supporting Information: Study Protocol
Time Frame: IPD will be shared after the study publication, for at least 5 years.
Access Criteria: The anonymized preprocessed behavioral data will be shared using an open access repository. Additional raw data access requests will be reviewed using an online form. Requestors will be required to sign a data access agreement.